CLINICAL TRIAL: NCT07115628
Title: Accelerated dTMS Treatment for ECT-non Responders
Brief Title: Accelerated TMS for Treatment-Resistant ECT
Acronym: A-TREC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Sara De Witte, PI, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-2024-380; Department of psychiatry (Other: UZ Brussel)
Record Dates: First submitted 2025-07-30; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder; MDD; Electroconvulsive therapy; ECT; Transcranial Magnetic Stimulation; TMS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TMS (Experimental): dTMS for depressed patients who did not improve after ECT. Patients will receive a 4-day course of active accelerated dTMS (Brainsway H1 coil; 20 sessions in total).
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — TMS is a non-invasive brain stimulation technique
  Other Names: TMS; adTMS

SUMMARY:
This study investigates whether an additional treatment using transcranial magnetic stimulation (TMS) can help severely depressed patients who did not respond well to electroconvulsive therapy (ECT).

All participants will first receive standard ECT treatment for depression, including brain scans (fMRI), psychological testing, clinical assessments, and the collection of blood and stool samples. If the ECT treatment is not effective, patients will be invited to participate in a second part of the study where they receive a 4-day course of accelerated TMS (20 sessions in total).

The study aims to assess whether this additional TMS treatment can reduce depressive symptoms. The study also explores how brain structure, genetics, and gut health may relate to treatment success. In total, 200 patients will be included.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is a well-established and effective treatment for severe major depressive disorder. However, a significant proportion of patients do not achieve remission after ECT, and effective follow-up treatment options for these non-responders remain limited.

This phase IV study explores the clinical effectiveness of an additional course of accelerated deep transcranial magnetic stimulation (dTMS) in patients who show partial or no response to ECT. The accelerated dTMS protocol consists of 20 sessions delivered over four consecutive days.

All patients initially undergo standard ECT treatment, accompanied by comprehensive psychological testing, clinical assessments, functional MRI scans (pre- and post-ECT), and collection of blood and stool samples. These data will be used to evaluate treatment response and investigate biological correlates of treatment outcomes, such as microbiome composition and genetic biomarkers.

Patients who do not reach remission after state-of-the-art ECT will be offered the opportunity to participate in the interventional phase of the study, receiving accelerated dTMS treatment, followed by a third fMRI scan and additional clinical, psychological testing, and biological sampling.

The primary goal is to assess whether this additional dTMS treatment improves remission rates. Secondary goals include evaluating brain-based, genetic, and gut-related predictors of treatment response, with the aim of guiding more personalized treatment strategies in the future.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder (MDD)
* Age between 18 - 70 years
* Referred for ECT treatment

Exclusion Criteria:

* A personal history of seizures or epilepsy, a history of seizures or epilepsy in first degree relatives and the presence of any known factor that can lower the seizure threshold (sleep deprivation, abuse substance, etc.), previous head injury and the presence of metallic implants in the cephalic region (e.g., aneurysm clips, shunts, stimulators, cochlear implants, electrodes) except dental fill-ings and the presence of cardiac pacemakers, neurostimulators, surgical clips or other electronic equipment, comorbidity with some neurological disorders: increased intracranial pressure, space-occupying lesion, history of stroke or transient ischemic attack, brain aneurysm and any structural brain damage with increased risk for epilepsy detected with MRI
* Patients with cognitive disturbances or dementia (Mini Mental State) < 24
* Suicide attempt within 6 months before the start of the study or pre-sent risk of suicide per the investigator's clinical judgment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Depression Severity - Clinician-Rated | Baseline (within 1 week before first ECT); within 1 week after last ECT session (variable duration); within 1 week after adTMS (20 sessions over 4 days; ECT non-responders only)
  Change in depressive symptom severity as measured by the 17-item Hamilton Depression Rating Scale (HDRS-17). Treatment response is defined as a ≥50% reduction in HDRS score from baseline. Remission is defined as an HDRS score ≤7.

SECONDARY OUTCOMES:
Change in Depression Severity - Self-Reported | Baseline (within 1 week before first ECT); within 1 week after last ECT session (variable duration); within 1 week after adTMS (20 sessions over 4 days; ECT non-responders only)
  Self-reported depressive symptoms measured using the Beck Depression Inventory-II (BDI-II)
Change in Suicidal Ideation - Clinician-Rated | Baseline (within 1 week before first ECT); within 1 week after last ECT session (variable duration); within 1 week after adTMS (20 sessions over 4 days; ECT non-responders only)
  Change in suicidal ideation evaluated using the Columbia-Suicide Severity Rating Scale (C-SSRS)
Psychological testing | Baseline (within 1 week before first ECT); within 1 week after last ECT session (variable duration); within 1 week after adTMS (20 sessions over 4 days; ECT non-responders only)
  Working memory task and psychomotor task
Neuroimaging | Baseline (within 1 week before first ECT); within 1 week after last ECT session (variable duration); within 1 week after adTMS (20 sessions over 4 days; ECT non-responders only)
  fMRI (functional and structural MRI) + emotion regulation task

OTHER OUTCOMES:
Gut Microbiome Composition | Baseline (within 1 week before first ECT); within 1 week after last ECT session (variable duration); within 1 week after adTMS (20 sessions over 4 days; ECT non-responders only)
  Analysis of gut microbiota composition using stool samples collected at three time points. The aim is to examine associations between microbial diversity/composition and clinical response to ECT and, in non-responders, to subsequent accelerated dTMS. Changes in microbial profiles will be compared between responders and non-responders to each treatment phase, to explore the predictive and modulatory role of the gut-brain axis in depression treatment outcomes.
Genetic and Epigenetic Biomarkers in Relation to Treatment Response | Baseline (within 1 week before first ECT); within 1 week after last ECT session (variable duration); within 1 week after adTMS (20 sessions over 4 days; ECT non-responders only)
  Genetic and epigenetic profiling will be performed on blood samples collected at multiple time points. The aim is to identify biological markers that predict or correlate with clinical response to ECT and, for non-responders, to accelerated dTMS. Differences in genetic and epigenetic profiles will be examined between responders and non-responders at each treatment phase to support the development of personalized treatment strategies for major depressive disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No